CLINICAL TRIAL: NCT02237248
Title: Functional Testing, and Biomechanics Before and After Scoliosis Surgery
Brief Title: Function and Scoliosis Surgery
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00055257
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent Idiopathic Scoliosis; Functional Movement Screen; Y Balance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to examine the changes in function and performance biomechanics in patients undergoing spinal fusion corrective surgery for adolescent idiopathic scoliosis (AIS).

DETAILED DESCRIPTION:
Methods will consist of movement studies, questionnaires, and chart review. The recruited subjects will be followed at the usual clinical schedule of pre-op, 6-week, 3 -, 6- and 12-month post-operative follow-up visits. After signing informed consent, age at time of surgery, height, weight, body composition, leg length will be recorded to be used during data processing. Chart review will further yield data on Cobb angle, Lenke Scoliosis classification, instrumentation used during surgery, and level of spinal fusion. All subjects will be asked to complete assessments of activity level (Marx Score, Tegner Activity Score), general health (EQ-5D), and a validated scoliosis survey (Scoliosis Research Study questionnaire SRS-22). Movement studies will consist of the Lower Quarter Y Balance Test (YBT-LQ), and Functional Movement Screen (FMS), and measures of forward flexion, right and left lateral bending, and right and left trunk rotation. These measures will be assessed preoperatively and at postoperative follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic scoliosis
* Patients identified to undergo spinal fusion surgery
* Treated at Duke University Medical Center

Exclusion Criteria:

* Neuromuscular or congenital scoliosis

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients that are undergoing spinal fusion surgery to treat idiopathic scoliosis.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Change in Lower Quarter Y-Balance Test (YBT-LQ) | Preoperatively; 6wks, 3mos, 6mos, and 12mos Postoperatively
  The YBT-LQ is a test of dynamic balance in unilateral stance that has been deemed to be reliable and valid. The YBT-LQ consists of each patient standing on one leg and reaching as far as they can with their non-stance leg in the anterior, posteromedial and posterolateral direction while standing on the other foot on a centralized stance platform.
Change in Functional Movement Screen (FMS) | Preoperatively; 6wks, 3mos, 6mos, and 12mos Postoperatively
  The FMS is a screening tool used to identify limitations or asymmetries in movement patterns by executing seven motions. Activities include a deep squat, lunges, hurdle steps, a push-up, straight-leg raises, shoulder mobility assessments, and rotary stability assessments.

SECONDARY OUTCOMES:
Change in Tegner Activity Scale | Preoperatively; 6wks, 3mos, 6mos, and 12mos Postoperatively
Change in Marx Activity Scale | Preoperatively; 6wks, 3mos, 6mos, and 12mos Postoperatively
Change in EQ-5D | Preoperatively; 6wks, 3mos, 6mos, and 12mos Postoperatively
Change in SRS-22 | Preoperatively; 6wks, 3mos, 6mos, and 12mos Postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Robert K Lark, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States